CLINICAL TRIAL: NCT03253731
Title: Interhemispheric Interaction of Parieto-Motor Cortico-Cortical Plasticity in Human Brain
Brief Title: Interhemispheric Interaction of Parieto-Motor Cortico-Cortical Plasticity
Status: Withdrawn | Type: Observational
Why Stopped: Investigator left the NIH.
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 170151; 17-N-0151
Record Dates: First submitted 2017-08-17; First posted 2017-08-18 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Healthy Volunteers
Keywords: Brain Plasticity; Healthy Volunteers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Healthy Volunteers: 15 healthy volunteers

SUMMARY:
Background:

The two hemispheres of the brain are connected. Changes in one hemisphere affect the other through this connection. Research has shown that training new skills in one hand improves the same skills for the other hand. Researchers want to learn more about how the brain works to transfer the skills to the other hand.

Objective:

To learn how changes on one side of the brain affect the other side. To study the activity of the left and right sides of the brain in healthy adults.

Eligibility:

Healthy volunteers ages 18-55 years old who are right-handed.

Design:

Participants will be screened with a medical history and physical exam. They will complete a questionnaire about their handedness. This may be done on paper or on a computer. Participants may have urine pregnancy tests.

Participants will have 2 study visits.

Participants will have a structural magnetic resonance imaging (MRI) scan. MRI uses a strong magnetic field and radio waves to take pictures of the brain. The scanner is a metal cylinder in a strong magnetic field. Participants will lie on a table that slides in and out of the cylinder.

Participants will have transcranial magnetic stimulation (TMS). Two wire coils will be placed on the scalp. A brief electrical current passes through the coil and creates a magnetic pulse that affects brain activity. Participants may be asked to tense certain muscles or do simple tasks during TMS.

Participants will have electromyography. Small sticky pad electrodes will be attached to the skin on the hands. Muscle activity will be recorded during the TMS procedure.

DETAILED DESCRIPTION:
Objective:

The purpose of this study is to evaluate the effect of long-term potentiation (LTP)-like cortical plasticity induced by parieto-motor cortico-cortical paired associative stimulation (cc-PAS) on the contralateral hemisphere and interhemispheric interactions in normal brain using dual-site transcranial magnetic stimulation (TMS). We will explore the ipsilateral and contralateral effects of cc-PAS over the left primary motor cortex (M1). We hypothesize that the motor evoked potential (MEP) at S50 (the motor evoked potential) will change after cc-PAS in the left hemisphere, which stimulates M1 after PPC (effective cc-PAS), not only on the right first dorsal interosseous (FDI) muscle, but also the left FDI muscle.

In addition, we hypothesize that the MEP at S50 will change after cc-PAS in the left hemisphere, which stimulates PPC after M1 (ineffective cc-PAS), on the right FDI muscle but not the left FDI muscle.

Study population

We intend to study 15 healthy-volunteers to have 12 who complete the study. Subjects will complete up to one screening visit and two study visits involving two intervention.

Design

Subjects will come for one screening visit and two outpatient study visits. The screening visit and the first study visit can be performed the same day. The second study visit will be done approximately 1 week after the first one. TMS-induced electromyographic (EMG) activity of hand muscles will be recorded as MEPs. Using single TMS measure on both the left and right M1, we will measure MEPs and input-out (I-O) curve for the right and left FDI muscle and abductor digiti minimi (ADM) muscle, respectively. Using a paired-pulse TMS paradigm, interhemispheric inhibition (IHI) from the left M1 to the right M1, short-interval intracortical inhibition (SICI) and intracortical facilitation (ICF) will be measured on the left FDI and ADM muscles. Then, the subjects will undergo two plasticity induction procedures of the parieto-motor cc-PAS sessions. One of those is the hypothesized efficacious cc-PAS session and the other one is the control, a hypothesized ineffective cc-PAS session. The two sessions will be separated by approximately one week. Each session consists of 100 pairs of double stimulation to the left PPC and left M1. MEPs, I-O curve on the bilateral M1, IHI from the left M1 to the right M1, SICI and ICF will be remeasured during the 60 min after receiving cc-PAS.

Outcome measures

Primary outcome:

The primary outcome measure will be MEP amplitude from the bilateral M1 with respect to time (before, immediately and 30-45 min after intervention) after induction of cc-PAS plasticity over the left hemisphere in each session. The amplitude of MEPs on each side of M1 will be compared between before and after cc-PAS with respect to time, using ANOVA in each session.

Secondary outcome:

The degree of IHI from the left M1 to the right M1, SICI and ICF with respect to time (before, immediately and 30-45 min after intervention) will be compared by the ANOVA test. The degree of IHI and the change of IHI will be correlated with the primary outcome as measured with a correlation analysis.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Between the age of 18 and 55 years
* Right-handed
* English speaking
* Ability to give informed consent

EXCLUSION CRITERIA:

* Illegal drugs use within the past 6 months based on history alone
* Abnormal findings on neurologic examination
* Have more than 7 alcoholic drinks a week in the case of a woman or 14 alcoholic drinks a week in the case of a man
* History of or current brain tumor, stroke, head trauma with loss of consciousness >few seconds, epilepsy or seizures
* History of or current episode of major depression or any major psychiatric illness (axis I disorders)
* Current diagnosis of neurologic disorder
* Presence of pacemaker, intracardiac lines, implanted pumps or stimulators, or metal objects inside the eye or skull. Dental fillings and dental braces are allowed.
* Open scalp wounds or scalp infection
* Employees and/or staff of HMCS/NINDS
* Taking benzodiazepines at the time of the entire study or within 12 days prior to the study. NOTE: Medication will not be stopped or held for participation in this study.
* Taking, at the time of the entire study or within 2 weeks prior to the study, any medication that acts as a central nervous system stimulant or that is known to lower seizure threshold, including, imipramine, amitriptyline, doxepin, nortriptyline, maprotiline, chlorpromazine, foscarnet, ganciclovir, ritonavir, amphetamines, ketamine, gamma-hydroxybutyrate (GHB), theophylline, mianserin, fluoxetine, fluvoxamine, paroxetine, sertraline, citalopram, reboxetine, venlafaxine, duloxetine, bupropion, mirtazapine, fluphenazine, pimozide, haloperidol, olanzapine, quetiapine, aripiprazole, ziprasidone, risperidone, chloroquine, mefloquine, imipenem, penicillin, ampicillin, cephalosporins, metronidazole, isoniazid, levofloxacin, cyclosporine, chlorambucil, vincristine, methotrexate, cytosine arabinoside, BCNU, lithium, antihistamines, and sympathomimetics. NOTE: Medication will not be stopped or help for participation in this study.
* Being pregnant
* You may not be eligible to have MRI or TMS in this study if:

  * You have metal in your body which would make having an MRI scan unsafe, such as pacemakers, stimulators, pumps, aneurysm clips, metallic prostheses, artificial heart valves, cochlear implants or shrapnel fragments, or if you were a welder or metal worker, since you may have small metal fragments in the eye.
  * You are uncomfortable in small closed spaces (you have claustrophobia) so that you would feel uncomfortable in the MRI machine.
  * You are not able to lie comfortably on your back for up to 1 hour
  * You have a hearing loss reported in the history or detected in the routine physical examination

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy Volunteers
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-08-11 (Actual); Primary Completion 2018-11-09 (Actual); Study Completion 2018-11-09 (Actual)

PRIMARY OUTCOMES:
MEP amplitude at S50 over each side of M1 with respect to time (before, and immediately after and 30-45 min after cc-PAS over the left M1). | 3 timepoints

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hallett, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)

REFERENCES:
- [Background] Awiszus F. TMS and threshold hunting. Suppl Clin Neurophysiol. 2003;56:13-23. doi: 10.1016/s1567-424x(09)70205-3. No abstract available. PMID 14677378
- [Background] Bloom JS, Hynd GW. The role of the corpus callosum in interhemispheric transfer of information: excitation or inhibition? Neuropsychol Rev. 2005 Jun;15(2):59-71. doi: 10.1007/s11065-005-6252-y. PMID 16211466
- [Background] Arai N, Muller-Dahlhaus F, Murakami T, Bliem B, Lu MK, Ugawa Y, Ziemann U. State-dependent and timing-dependent bidirectional associative plasticity in the human SMA-M1 network. J Neurosci. 2011 Oct 26;31(43):15376-83. doi: 10.1523/JNEUROSCI.2271-11.2011. PMID 22031883